CLINICAL TRIAL: NCT01295762
Title: Immunomonitoring of Children With Neuroblastoma for the Development of Antitumor Immunotherapy Strategies
Brief Title: Immunomonitoring of Children With Neuroblastoma
Acronym: Immuneuro
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IMMUNEURO
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Neuroblastoma
Keywords: Children; Cancer; Immunomonitoring; Prognostic/Predictive Factors; Immunotherapy
MeSH Terms: conditions — Neuroblastoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Type of neuroblastoma (Other): Neonatal stages I Localized immediately resectable stages Localized immediately unresectable stages High-risk neuroblastoma Relapsed neuroblastoma
  Interventions: Other: Immunological analyses

INTERVENTIONS:
Other: Immunological analyses — Immunological analyses will be done on blood, bone marrow and tumor samples, at diagnosis, and during the treatment of children diagnosed for neuroblastoma (up to 3 time points). These types of samples are routinely done during conventional neuroblastoma treatment.
  Other Names: No intervention other names

SUMMARY:
Apart from brain tumors, Neuroblastoma is the most common solid tumor during childhood. About 50% of the cases present at diagnosis with factors of bad prognosis. During the last two decades, despite increased therapeutic intensity during induction and consolidation of high-risk neuroblastomas, the 5 year overall survival of high risk neuroblastoma remains in between 30 to 40% depending on studies.

Besides strategies of high-dose chemotherapy followed by autologous transplantation of hematopoietic stem cells, and differentiating molecules (retinoids), immunotherapy will become one of the leading anti-neuroblastoma targeted therapy. No therapeutic strategies or molecules obtained such gains of survival ever before.

Studying the immune system of children with neuroblastoma at diagnosis and during their treatment will help us to determine when we should test active or passive immunotherapy strategies. Moreover, this study would allow us to specify the cause of tumor immune tolerance in neuroblastoma, on which we have few data in comparison to adult tumors.

This will be a multicentric, pilot, prospective, open, study that will not require unusual diagnostic interventions. This study will be transversal (all neuroblastoma stages included) in order to determine comparative criteria between low and high risk neuroblastoma. It will also be longitudinal (from diagnosis to post-treatment follow-up) in order to specify evolutionary aspects of immunity under radio-chemotherapy and retinoic acid therapy.

Immunological analyses will be done on blood, bone marrow and tumor samples, at diagnosis, and during the treatment of children diagnosed for neuroblastoma (up to 3 time points). These types of samples are routinely done during conventional neuroblastoma treatment.

DETAILED DESCRIPTION:
The main objective of the study is the description of immune effectors in the blood, marrow and tumor diagnosis.

During 3 years, this trial will include 30 children from pediatric oncology units of Lyon, Saint-Etienne, Grenoble and Clermont-Ferrand.

The study duration is 5 years. Children follow-up scheduled for at least 2 years in order to determine predictive factors of therapeutic efficiency and survival.

Multi-parametric marker sets (6-8 markers per sample) have already developed and validated for analyzing the absolute amount and proportion of immune subpopulations (B, TCD4+, TCD8+, Treg, NK, DC) and activation status (PD1, ICOS, CD39, CD73, CD62L, CCR7, CD45RO, CD45RA, CD86, Ox40, CD137, CTLA4) on a small volume. At least, these analyses will be performed on each blood and marrow sample. If the amount of blood and mononuclear cells harvested allows it, functional analyses will be undertaken (intracytoplasmic cytokines in response to activation for T, DC, NK; protocols been set up).

Immunostainings will be performed on tumor samples at diagnosis and after resection of the primary tumor, in order to determine the expression and evolution of several immunomodulatory molecules on neuroblastoma cells (HLA class I & II, HLA-G, IDO, IL10,…)., and also determine the immune infiltrate within the tumor microenvironment (lymphocytes Treg, cellules dendritiques, MDSC,…). The techniques used will mostly be those of classical immunology (IHC, IF, FACS), and have already been set-up in our INSERM team for adult tumors.

Children's plasma will be screened for specific anti-tumor immunoglobulins at diagnosis and at key treatment time points. In the meanwhile, levels of circulating cytokines concentrations will be evaluated by Luminex, especially those known to have inhibitory effects on immune effectors: IL-4, IL-5, IL-6, IL-10, TGF-beta, HLA-Gs, TNF-alpha, IFN-gama, IL-2, IL-12, IL-27, IL-17 and CD40L (already in place).

ELIGIBILITY:
Inclusion Criteria:

* Age <= 21 years
* Patient with neuroblastoma any stage, in the first line or relapsed, or suspicion of neuroblastoma
* Covered by a medical insurance
* Written, signed informed consent (patient, and parents if minor child)

Exclusion Criteria:

* Patients who received corticosteroids within 15 days prior to sampling
* Patients receiving immunosuppressive therapy
* Chemotherapy before sampling began
* Neuroblastoma in a genetic syndrome predisposing
* Deterioration of clinical status

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Description of immune effectors in the blood, marrow and tumor diagnosis. | 1 year
  Rate effectors immunitaires in blood, marrow and tumor present at diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien MARABELLE, MD, Principal Investigator — IHOP
Locations (4):
- France (4):
  - Hopital D'Estaing, Clermont-Ferrand
  - Chu Grenoble - Hopital Nord, La Tronche
  - IHOP, Lyon
  - Chu - Hopital Nord, Saint-Priest-en-Jarez

REFERENCES:
- [Result] Marabelle A, Merlin E, Halle P, Paillard C, Berger M, Tchirkov A, Rousseau R, Leverger G, Piguet C, Stephan JL, Demeocq F, Kanold J. CD34+ immunoselection of autologous grafts for the treatment of high-risk neuroblastoma. Pediatr Blood Cancer. 2011 Jan;56(1):134-42. doi: 10.1002/pbc.22840. PMID 21058288
- [Result] Bertrand A, Marec-Berard P, Raverot G, Trouillas J, Marabelle A. Cabergoline therapy of paraneoplastic Cushing syndrome in children. Pediatr Blood Cancer. 2010 Sep;55(3):589-90. doi: 10.1002/pbc.22581. No abstract available. PMID 20658641
- [Result] Marabelle A, Bergeron C, Billaud G, Mekki Y, Girard S. Hemophagocytic syndrome revealing primary HHV-6 infection. J Pediatr. 2010 Sep;157(3):511. doi: 10.1016/j.jpeds.2010.02.064. Epub 2010 Apr 18. No abstract available. PMID 20400100
- [Result] Marabelle A, Sapin V, Rousseau R, Periquet B, Demeocq F, Kanold J. Hypercalcemia and 13-cis-retinoic acid in post-consolidation therapy of neuroblastoma. Pediatr Blood Cancer. 2009 Feb;52(2):280-3. doi: 10.1002/pbc.21768. PMID 18839433
- [Result] Marabelle A, Campagne D, Dechelotte P, Chipponi J, Demeocq F, Kanold J. Focal nodular hyperplasia of the liver in patients previously treated for pediatric neoplastic diseases. J Pediatr Hematol Oncol. 2008 Jul;30(7):546-9. doi: 10.1097/MPH.0b013e3181691709. PMID 18797204
- [Result] Kanold J, Paillard C, Tchirkov A, Merlin E, Marabelle A, Lutz P, Rousseau R, Baldomero H, Demeocq F. Allogeneic or haploidentical HSCT for refractory or relapsed solid tumors in children: toward a neuroblastoma model. Bone Marrow Transplant. 2008 Oct;42 Suppl 2:S25-30. doi: 10.1038/bmt.2008.279. PMID 18978740
- [Result] Kanold J, Merlin E, Halle P, Paillard C, Marabelle A, Rapatel C, Evrard B, Berger C, Stephan JL, Galambrun C, Piguet C, D'Incan M, Bordigoni P, Demeocq F. Photopheresis in pediatric graft-versus-host disease after allogeneic marrow transplantation: clinical practice guidelines based on field experience and review of the literature. Transfusion. 2007 Dec;47(12):2276-89. doi: 10.1111/j.1537-2995.2007.01469.x. Epub 2007 Aug 30. PMID 17764513